CLINICAL TRIAL: NCT01348087
Title: An Open-label Study to Evaluate the Long-term Safety, Tolerability and Efficacy of AFQ056 in Adult Patients With Fragile X Syndrome
Brief Title: Long-term, Safety, Tolerability and Efficacy Study of AFQ056 in Adult Patients With Fragile X Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study treatment AFQ056 failed to demonstrate efficacy in the adult patient with Fragile X Syndrome in 2 other clinical studies (CAFQ056B2214 and CAFQ056A2212)
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAFQ056B2279; 2011-001952-12 (EudraCT Number)
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome; Martin-Bell Syndrome; Genetic Diseases; X-Linked; Escalante's syndrome
MeSH Terms: conditions — Fragile X Syndrome; Genetic Diseases, Inborn | interventions — mavoglurant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AFQ056 100 mg (Bid) (Experimental): All patients initiated treatment with AFQ056 at a starting dose of 25 milligram (mg) twice daily. The dose was titrated from 25mg bid to 50mg bid, 75mg bid and 100mg bid at weekly intervals. Dose adjustments (up- and down titrations) were permitted as needed to manage any tolerability issues and to ensure that patients reach their highest tolerated dose not to exceed 100mg bid.
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056 — The investigational drug, AFQ056, will be provided as hard gelatin capsules. Two different oral dosage strengths, identical in appearance, will be used.

SUMMARY:
The purpose of this study is to generate long-term safety, tolerability and efficacy data for AFQ056 in eligible adult patients with FXS who have participated in the CAFQ056A2212 (NCT01253629).study and patients who have participated in the previous proof-of-concept study CAFQ056A2204 (NCT00718341).

DETAILED DESCRIPTION:
A 148 patients were enrolled into this treatment extension trial conducted for at least 3 years. This extension trial was terminated after the decision to terminate the AFQ056 development program. The decision was based on the results of two randomized, double blind, placebo controlled phase IIb trials in adult and adolescent FXS patients (CAFQ056A2212 and CAFQ056B2214respectivly), both of which failed to demonstrate efficacy in the FXS population. As this extension trial was terminated, only the primary objective and safety are represented.

ELIGIBILITY:
Inclusion criteria Group 1 patients

* Had to have completed the CAFQ056A2212 study or another study of AFQ056 which included adult FXS patients within one week of enrollment into the open-label study.
* Females of child-bearing potential had to follow protocol requirements with respect to contraception.
* Have a caregiver or caregivers who spent, on average, at least six hours per day with the patient, who were willing and capable of supervising treatment, providing input into efficacy and safety assessments, and accompanying the patient to study visits.

Group 2:

* Had to have:
* Completed Study CAFQ056A2204.
* Completed Study CAFQ056A2212 or another study of AFQ056 which included adult patients with FXS but enrollment into the current study was delayed for more than a week.
* Discontinued prematurely from Study CAFQ056A2212 or another study of AFQ056 which included adult patients with FXS due to intolerability of the dosage in the patient's assigned treatment group.
* Females of child-bearing potential had to follow protocol requirements with respect to contraception.
* Have a caregiver or caregivers who spent, on average, at least six hours per day with the patient, who were willing and capable of supervising treatment, providing input into efficacy and safety assessments, and accompanying the patient to study visits

Exclusion criteria

Any advanced, severe or unstable disease

* History of severe self- injurious behavior
* History of uncontrolled seizure disorder or resistant to therapy within the past 2 years (Patients who are clinically stable under anti-convulsant therapy for the past 2 years are not excluded)
* History of clinically significant allergies requiring hospitalization or non- inhaled corticosteroid therapy (asthma, anaphylaxis, etc.)
* Using (or used within 6 weeks before baseline) concomitant medications that are potent inhibitors or inducers of CYP3A4
* Using glutamatergic agents (riluzole, memantine, etc.) or lithium, digoxin, or warfarin within 6 weeks of baseline Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (10):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Staten Island, New York
  - Novartis Investigative Site, Media, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
- Australia (3):
  - Novartis Investigative Site, Ryde, New South Wales
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Caulfield, Victoria
- Canada (2):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Sherbrooke, Quebec
- Novartis Investigative Site, Glostrup Municipality, Denmark
- France (2):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Paris
- Germany (4):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Genova, GE, Italy
- Spain (2):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Edinburgh, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 centers in 10 countries
Pre-assignment Details: A total of 148 patients were enrolled and treated, including 1 patient who discontinued and was later re-enrolled under a new patient number. Category 1 patients received AFQ056 in the core study and enrolled in the extension within 7 days of completing the core study; Category 2 included all other patients enrolled into the extension study
Groups:
- AFQ056 Total: Participants from a previous AFQ056 study who entered the open-label extension study were administered AFQ056 capsules at a starting dose of 25 milligram (mg) twice daily (bid) and then titrated to 50 mg bid, 75 mg bid and 100 mg bid at weekly intervals
Period: Overall Study
Arm/Group | AFQ056 Total
Started | 148
Completed | 0
Not Completed | 148
Not completed — Unsatisfactory therapeutic effect | 35
Not completed — Administrative problems | 79
Not completed — protocol deviation | 1
Not completed — Lost to Follow-up | 1
Not completed — Subject withdrew consent | 7
Not completed — Adverse Event | 25

BASELINE CHARACTERISTICS:
Groups:
- AFQ056: Participants from a previous AFQ056 study who entered the open-label extension study were administered AFQ056 capsules at a starting dose of 25 milligram (mg) twice daily (bid) and then titrated to 50 mg bid, 75 mg bid and 100 mg bid at weekly intervals
Arm/Group | AFQ056
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.6 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 138

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs).
Description: Adverse events were summarized for the open-label treatment period, where the open-label treatment period is defined based on how AEs were collected and reported according to the manner in which patients entered the current study and which treatment (AFQ056 or placebo) they were receiving in the previous study. AEs which were continuing from the core study or that started after the end of core study but prior to first dose of open-label study medication in the extension study for Category 1 patients are shown under ('Prior to Ext. first dose'). AEs which started during the open-label treatment period are presented based on the last AFQ056 dose taken on or before the onset date of the AE (25 mg bid; 50 mg bid; 75 mg bid; or 100 mg bid). No efficacy data presented as study was terminated
Time Frame: Prior to first dose in extension study, Baseline (start of study treatment in extension study) to End of trial
Population: The analysis was performed in the safety set (SS) population, defined as participants who received at least one dose of study medication and had at least one safety assessment occurring after first dose of extension study medication. Here, 'Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure
Measure: Number; unit: Participants
Arm/Group | Prior to Ext First Dose | AFQ056 25mg Bid | AFQ056 50mg Bid | AFQ056 75mg Bid | AFQ056 100mg Bid | AFQ056 Total
Number analyzed (Participants) | 40 | 147 | 148 | 141 | 135 | 148
Participants
  At least one AE | 9 | 49 | 47 | 50 | 112 | 138
  At least one severe AE | 1 | 1 | 2 | 5 | 18 | 24
  Any serious or significant AE | 0 | 1 | 0 | 1 | 6 | 7
  SAE | 0 | 1 | 0 | 1 | 6 | 7
  Discontinued due to SAE | 0 | 1 | 0 | 1 | 1 | 3
  Discontinued due to non serious AE | 0 | 4 | 5 | 4 | 11 | 22

ADVERSE EVENTS:
Groups:
- Prior to Ext.First Dose: Prior to Ext.first dose
- AFQ056 25 mg Bid: AFQ056 25 mg bid
- AFQ056 50 mg Bid: AFQ056 50 mg bid
- AFQ056 75 mg Bid: AFQ056 75 mg bid
- AFQ056 100 mg Bid: AFQ056 100 mg bid
Arm/Group | Prior to Ext.First Dose | AFQ056 25 mg Bid | AFQ056 50 mg Bid | AFQ056 75 mg Bid | AFQ056 100 mg Bid | AFQ056 Total
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/147 | 0/148 | 1/141 | 6/135 | 7/148
Other Adverse Events (participants affected / at risk) | 6/40 | 26/147 | 28/148 | 36/141 | 88/135 | 117/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior to Ext.First Dose (N=40) | AFQ056 25 mg Bid (N=147) | AFQ056 50 mg Bid (N=148) | AFQ056 75 mg Bid (N=141) | AFQ056 100 mg Bid (N=135) | AFQ056 Total (N=148)
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 3
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 2
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior to Ext.First Dose (N=40) | AFQ056 25 mg Bid (N=147) | AFQ056 50 mg Bid (N=148) | AFQ056 75 mg Bid (N=141) | AFQ056 100 mg Bid (N=135) | AFQ056 Total (N=148)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 7 | 10
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 14 | 18
Asthenia (General disorders) | 0 | 1 | 0 | 5 | 8 | 9
Fatigue (General disorders) | 0 | 1 | 2 | 3 | 3 | 9
Nasopharyngitis (Infections and infestations) | 3 | 2 | 4 | 3 | 21 | 27
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 1 | 3 | 16 | 24
Dizziness (Nervous system disorders) | 1 | 5 | 4 | 1 | 5 | 13
Headache (Nervous system disorders) | 0 | 4 | 3 | 7 | 14 | 21
Aggression (Psychiatric disorders) | 0 | 6 | 8 | 5 | 11 | 22
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 3 | 10 | 13
Anxiety (Psychiatric disorders) | 0 | 1 | 3 | 3 | 10 | 16
Insomnia (Psychiatric disorders) | 1 | 4 | 3 | 7 | 12 | 23
Irritability (Psychiatric disorders) | 1 | 0 | 7 | 4 | 6 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 2 | 9 | 16

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate this study prematurely, as the study treatment failed to demonstrate efficacy in target population in two other clinical studies: CAFQ056B2214 (NCT01357239) and CAFQ056A2212 (NCT01253629).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety